CLINICAL TRIAL: NCT05687253
Title: A Phase 2, Randomized, Double-Blind, Active-Controlled, Evaluation of Intubation Conditions Following BX1000 or Rocuronium in Subjects Undergoing Surgery
Brief Title: Evaluation of Intubation Conditions Following BX1000 or Rocuronium in Subjects Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDX-22-006
Record Dates: First submitted 2022-12-09; First posted 2023-01-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neuromuscular Blockade; Anesthesia; Surgery
Keywords: Intubation
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, active controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BX1000 0.15 mg/kg (Experimental): BX1000 0.15 mg/kg IV Bolus
  Interventions: Drug: BX1000
- BX1000 0.25 mg/kg (Experimental): BX1000 0.25 mg/kg IV Bolus
  Interventions: Drug: BX1000
- BX1000 0.35 mg/kg (Experimental): BX1000 0.35 mg/kg IV Bolus
  Interventions: Drug: BX1000
- Rocuronium 0.6 mg/kg (Active Comparator): Rocuronium bromide 0.6 mg/kg IV Bolus
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: BX1000 — IV BX1000
  Arms: BX1000 0.15 mg/kg; BX1000 0.25 mg/kg; BX1000 0.35 mg/kg
Drug: Rocuronium Bromide — IV Rocuronium
  Arms: Rocuronium 0.6 mg/kg

SUMMARY:
Assessment of Intubation conditions following administration of neuromuscular blocking agents; BX1000 (investigational) or rocuronium (active control).

DETAILED DESCRIPTION:
Intubation conditions will be assessed in anesthetized subjects undergoing an elective surgical procedure utilizing general anesthesia. Following administration of IV anesthesia, subjects will have electromyography (EMG) neuromuscular monitoring device applied prior to administration of neuromuscular blocking agent (NMBA). NMBA will be administered and assessment of intubation conditions will begin 60 seconds after administration according to the methods defined in Viby-Mogensen 1996; assessment will be repeated at 90 and 120 seconds after administration when intubation has not already been completed.

After intubation is completed, subjects will progress to have their elective surgery completed and will be maintained under general anesthesia until neuromuscular function is recovered. Once recovered from anesthesia and extubation, subjects will be monitored in a recovery area until they are suitable to be discharged to the inpatient floor, after which time they may be discharged at the clinical discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent
* Undergoing elective surgery utilizing IV general anesthesia
* Normal airway assessment

Exclusion Criteria:

* Unstable disease or emergency surgical conditions
* Known hypersensitivity to rocuronium, other NMB or study medications
* History of anaphylaxis
* History of neuromuscular junction disease
* Personal or family history of malignant hyperthermia or pseudocholinesterase deficiency
* Diagnosed or suspected sleep apnea
* History of prior anesthetic complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Intubation Conditions | Within 2 minutes after administration
  Assessment of Intubation Conditions (Poor, Good, Excellent) Following Administration of Neuromuscular Blocking agent

SECONDARY OUTCOMES:
Assessment of Safety And Tolerability - Adverse Events | Within 30 days after administration
  Assessment of Incidence of Adverse Events Following Administration of Neuromuscular Blocking agent
Assessment of Safety And Tolerability - Blood Pressure | Within 30 days after administration
  Assessment of Changes in Blood Pressure Following Administration of Neuromuscular Blocking agent
Assessment of Safety And Tolerability - Heart Rate | Within 30 days after administration
  Assessment of Changes in Heart Rate Following Administration of Neuromuscular Blocking agent
Assessment of Safety And Tolerability - Blood Oxygen Saturation | Within 30 days after administration
  Assessment of Changes in Vital signs Following Administration of Neuromuscular Blocking agent
Assessment of Onset of Neuromuscular Blockade | Within 1 day after administration
  Measurement of Twitch Suppression via Electromyography Following Administration of Neuromuscular Blocking agent
Assessment of Neuromuscular Recovery | Within 1 day after administration
  Measurement of Twitch Recovery via Electromyography Following Administration of Neuromuscular Blocking agent

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Center, San Antonio, Texas
  - Research Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No